CLINICAL TRIAL: NCT01175746
Title: The Effect of Nicardipine on Kidney Function During Orthognathic Surgery Under Hypotensive Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3-2009-0196
Record Dates: First submitted 2010-08-02; First posted 2010-08-05 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Subjects
Keywords: healthy adult patients; ASA class I; hypotensive anesthesia
MeSH Terms: interventions — Nicardipine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nicardipine (Experimental)
  Interventions: Drug: Nicardipine
- remifentanil (Active Comparator)
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: Nicardipine
  Arms: nicardipine
Drug: remifentanil — 0.1-0.5 ugkg/min during hypotensive anesthesia
  Other Names: ultiva®
  Arms: remifentanil

SUMMARY:
Since nicardipine is known to protect kidney function, nicardipine infusion will result in better renal parameters measured in this study.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult patients undergoing hypotensive anesthesia

Exclusion Criteria:

* patients with any co-morbidity

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Creatinine Clearance | 2hr after the start of hypotensive anesthesia
  Hypotensive anesthesia means that we maintain the mean blood pressure between 55 & 65 mmHg during surgery to decrease the blood loss.
  The specific time point is exactly 2hr after we star to lower the blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Kim, Principal Investigator — Severance hospital, YUHS